CLINICAL TRIAL: NCT01634464
Title: The Role of Nutrition and Maternal Genetics on the Programming of Development of Fetal Adipose Tissue. Search for Markers of the Obesity Risk in Early Stages of Life
Brief Title: Role of Nutrition and Maternal Genetics on the Programming of Development of Fetal Adipose Tissue
Acronym: PREOBE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Abbott (Industry); Scottish Government NuGO EU Project (Unknown); University of Barcelona (Other); ICTAN-CSIC - Madrid - Spain (Unknown); Ludwig-Maximilians - University of Munich (Other); University of Nottingham (Other); University of Aberdeen (Other); Andalusian Agency of Knowledge (Other Government)
Responsible Party: Principal Investigator, Cristina Campoy, Professor, Universidad de Granada
Other Study IDs: P06-CTS-02341; 334602 Preobe Follow Up (Other Grant/Funding Number: Abbot Laboratories SA/General Foundation University of Granada - Enterprise)
Record Dates: First submitted 2012-03-19; First posted 2012-07-06 (Estimated); Last update posted 2012-07-09 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood and blood from the umbilical cord, serum, plasma, placental tissue, placental tissue treated with RNAlater, saliva, oral mucosa, urine, faeces, human milk
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Control group: women with 18.5 > BMI < 25
- Pregnant women with overweight: BMI≥25 before the pregnancy
- Pregnant women with obesity: BMI≥30 before the pregnancy
- Pregnant women with gestational diabetes: Gestational diabetes

SUMMARY:
In the PREOBE projects it is aimed to obtain genetic and biochemical biomarkers for the programming of obesity in early stages of life. This can be achieved by studying pregnant women with normal weight, overweight, obesity and gestational diabetes, and by analyzing how these conditions could impact on fetal growth and development; the risk of obesity in the offspring during the first 3 years of life will be also assessed (genetic polymorphisms of the most recognized genes related to obesity; gene expression of placental biomarkers indicators of early programming, polyunsaturated fatty acids, immunological and pro-inflammatory markers, analysis of endogenous and exogenous lipid peroxidation, allergies & neurodevelopmental assessment...). Moreover, the interaction of pathological maternal conditions with confounder factors that could have a role in the proposed outcomes will be also studied (maternal and child dietary intake, medical history and socioeconomic & environmental factors).

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women aged between 18 and 42
* singleton pregnancies
* pregnancy stage at recruitment: 12 weeks of pregnancy

Exclusion Criteria:

* Women who wish to participate in the study should not simultaneously participate in other research studies.
* Must be completely enclosed in one of the study of the groups without any possibility to be simultaneously incorporated on more groups of the study
* Mothers which are receiving any drug treatment, folate more than the 3rd first months, or DHA +/- vitamin supplements during pregnancy.
* Mothers affected by any disease other than those referred to the inclusion criteria, such hypertension or pre-eclampsia, foetal IUGR, mother infection during pregnancy, hypothyroidism / hyperthyroidism, hepatic diseases, renal disease,…
* Mothers following an extravagant diet or vegan diet.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 350 pregnant women aged between 18 and 42, with singleton pregnancies, were recruited at 12 weeks of pregnancy at the Clinical University Hospital 'San Cecilio' and "Mother-Infant" Hospital in the city of Granada, Spain
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2007-03; Primary Completion 2010-10 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Long-term evidence of early human programming of obesity measured by nutritional biomarkers, and the offspring growth and development. | Participants will be followed for the duration of the study, an expected average of 6 years
Long-term evidence of early human programming of obesity measured by genetic biomarkers, and the offspring growth and development. | Participants will be followed for the duration of the study, an expected average of 6 years
Long-term evidence of early human programming of obesity measured biochemical perinatal biomarkers, and the offspring growth and development. | Participants will be followed for the duration of the study, an expected average of 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Campoy, Professor, MD, Study Director — Universidad de Granada
Locations (1):
- Department of Pediatrics, School of Medicine, University of Granada, Granada, Spain

REFERENCES:
- [Result] Santacruz A, Collado MC, Garcia-Valdes L, Segura MT, Martin-Lagos JA, Anjos T, Marti-Romero M, Lopez RM, Florido J, Campoy C, Sanz Y. Gut microbiota composition is associated with body weight, weight gain and biochemical parameters in pregnant women. Br J Nutr. 2010 Jul;104(1):83-92. doi: 10.1017/S0007114510000176. Epub 2010 Mar 8. PMID 20205964
- [Result] Campoy C, Martin-Bautista E, Garcia-Valdes L, Florido J, Agil A, Lorente JA, Marcos A, Lopez-Sabater MC, Miranda-Leon T, Sanz Y, Molina-Font JA; grupo PREOBE. [Study of maternal nutrition and genetic on the foetal adiposity programming (The PREOBE study)]. Nutr Hosp. 2008 Nov-Dec;23(6):584-90. Spanish. PMID 19132267
- [Derived] Cerdo T, Ruiz-Rodriguez A, Acuna I, Torres-Espinola FJ, Menchen-Marquez S, Gamiz F, Gallo M, Jehmlich N, Haange SB, von Bergen M, Campoy C, Suarez A. Infant gut microbiota contributes to cognitive performance in mice. Cell Host Microbe. 2023 Dec 13;31(12):1974-1988.e4. doi: 10.1016/j.chom.2023.11.004. Epub 2023 Dec 4. PMID 38052208
- [Derived] Berglund SK, Garcia-Valdes L, Torres-Espinola FJ, Segura MT, Martinez-Zaldivar C, Aguilar MJ, Agil A, Lorente JA, Florido J, Padilla C, Altmae S, Marcos A, Lopez-Sabater MC, Campoy C; PREOBE team. Maternal, fetal and perinatal alterations associated with obesity, overweight and gestational diabetes: an observational cohort study (PREOBE). BMC Public Health. 2016 Mar 1;16:207. doi: 10.1186/s12889-016-2809-3. PMID 26931143
- [Derived] Torres-Espinola FJ, Berglund SK, Garcia-Valdes LM, Segura MT, Jerez A, Campos D, Moreno-Torres R, Rueda R, Catena A, Perez-Garcia M, Campoy C; PREOBE team. Maternal Obesity, Overweight and Gestational Diabetes Affect the Offspring Neurodevelopment at 6 and 18 Months of Age--A Follow Up from the PREOBE Cohort. PLoS One. 2015 Jul 24;10(7):e0133010. doi: 10.1371/journal.pone.0133010. eCollection 2015. PMID 26208217
- [Derived] Torres-Espinola FJ, Altmae S, Segura MT, Jerez A, Anjos T, Chisaguano M, Carmen Lopez-Sabater M, Entrala C, Alvarez JC, Agil A, Florido J, Catena A, Perez-Garcia M, Campoy C. Maternal PPARG Pro12Ala polymorphism is associated with infant's neurodevelopmental outcomes at 18 months of age. Early Hum Dev. 2015 Aug;91(8):457-62. doi: 10.1016/j.earlhumdev.2015.05.001. Epub 2015 May 26. PMID 26025336
- [Derived] Uhl O, Demmelmair H, Segura MT, Florido J, Rueda R, Campoy C, Koletzko B. Effects of obesity and gestational diabetes mellitus on placental phospholipids. Diabetes Res Clin Pract. 2015 Aug;109(2):364-71. doi: 10.1016/j.diabres.2015.05.032. Epub 2015 May 16. PMID 26021978